CLINICAL TRIAL: NCT00747058
Title: A Double Blind (3rd Party Open), Randomized, Placebo Controlled, Dose Escalating Study To Investigate The Safety, Toleration And Pharmacokinetics Of Single Oral Doses Of PF-03864086 In Healthy Male Subjects
Brief Title: A Study To Investigate The Safety, Toleration And Pharmacokinetics Of Single Oral Doses Of PF-03864086 In Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B0361006
Record Dates: First submitted 2008-08-18; First posted 2008-09-04 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Pain
Keywords: phase 1, human study, healthy volunteers
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy volunteers (Experimental)
  Interventions: Drug: PF-3864086
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-3864086 — The dosage form is POS (powdered oral suspension). Each subject will have 5 periods and the frequency (and duration) is once per period. The doses have been left flexible within the protocol but are listed as: 3, 10, 30, 60, 120, 240, 480 and 720 mg with an option to insert an additional dose cohort as well.
  Arms: healthy volunteers
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of PF-03864086 in healthy male human volunteers. Determine the pharmacokinetics (calculations of the rate of elimination of PF-03864086 from the body once the compound is ingested).

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers
* no drug history
* no other medication for 28 pre-dose

Exclusion Criteria:

* age below 21 years
* age above 55 years

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | measured intensively in the first 48 hours and continue out to day 14
Tolerability | measured intensively in the first 48 hours and continue out to day 14

SECONDARY OUTCOMES:
Temperature change | continuous recording over the first 48h post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0361006&StudyName=A%20Study%20To%20Investigate%20The%20Safety%2C%20Toleration%20And%20Pharmacokinetics%20Of%20Single%20Oral%20Doses%20Of%20PF-03864086%20In%20Healthy%20Male%20Subjects%0A